CLINICAL TRIAL: NCT01007656
Title: A Multiple-Dose Research Study on Safety Evaluation of the GD Antrodia Camphorata in 30 Healthy Adult Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Golden Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: IRC01080923
Record Dates: First submitted 2009-10-30; First posted 2009-11-04 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: healthy adult subjects; safety evaluation; GD Antrodia camphorata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GD Antrodia camphorata (Experimental): GD Antrodia Camphorata is the extract from mycelium of the fungus "Antrodia Camphorata" which is an endemic species in Taiwan. According to the literatures, mycelium of Antrodia camphorata is beneficial to health. Moreover, the study product GD Antrodia Camphorata has been approved by Department of Health, Taiwan as a health supplement (approval number A00124).
  Interventions: Dietary Supplement: GD Antrodia camphorata

INTERVENTIONS:
Dietary Supplement: GD Antrodia camphorata — Three 500mg capsules per oral dose, twice daily with an interval of 12 hours for 90 days

SUMMARY:
* Study design is multiple-dose, open-label study
* The purpose of this study is to evaluate the safety after twice daily GD Antrodia camphorata administration for 90 days in 30 healthy adult subjects.

  * Primary objective: The mean change from baseline in laboratory assessment after twice daily GD Antrodia camphorata administration at 90th day in 30 healthy adult subjects.
  * Secondary objective: The mean change from baseline in laboratory assessment after twice daily GD Antrodia camphorata administration at 10th, 20th, 30th, 45th and 60th day in 30 healthy adult subjects.
* Safety Measurement:

  * including SGOT(AST), SGPT(ALT), albumin, glucose, creatinine, uric acid, cholesterol, TG, r-GT, alkaline phosphatase, total bilirubin, D-Bil, BUN, TP, GLO will be documented at 1st, 10th, 20th, 30th, 45th, 60th and 90th day.
  * vital signs (heart rate, blood pressure, and body temperature) will be documented at 1st, 10th, 20th, 30th, 45th, 60th and 90th day.
  * Subjects will be monitored throughout the confinement portion of the study.

DETAILED DESCRIPTION:
* Study design is multiple-dose, open-label study
* Antrodia camphorata has been proved to alleviate liver injury and fibrosis induced by chemical and reduces ALT and AST according to the literatures.
* "GD Antrodia camphorata" will be marketed as dietary supplement.
* The purpose of this study is to evaluate the safety after twice daily GD Antrodia camphorata administration for 90 days in 30 healthy adult subjects.

  * Primary objective: The mean change from baseline in laboratory assessment after twice daily GD Antrodia camphorata administration at 90th day in 30 healthy adult subjects.
  * Secondary objective: The mean change from baseline in laboratory assessment after twice daily GD Antrodia camphorata administration at 10th, 20th, 30th, 45th and 60th day in 30 healthy adult subjects.
* Study design is multiple-dose, open-label study
* The study site is Pingtung Christian Hospital Ruiguang Branch.
* Safety Measurement:

  * including SGOT(AST), SGPT(ALT), albumin, glucose, creatinine, uric acid, cholesterol, TG, r-GT, alkaline phosphatase, total bilirubin, D-Bil, BUN, TP, GLO will be documented at 1st, 10th, 20th, 30th, 45th, 60th and 90th day.
  * vital signs (heart rate, blood pressure, and body temperature) will be documented at 1st, 10th, 20th, 30th, 45th, 60th and 90th day.
  * Subjects will be monitored throughout the confinement portion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult, aged between 20 to 40 years old
* Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, laboratory tests, chest X-ray and electrocardiogram
* The normal range of the body mass index should between 18.5 and 24.9; body mass equals [weight(Kg)]/[height(m)]2
* Normal laboratory determinations results (within normal range or considered not clinically significant by the investigator) including: SGOT (AST), SGPT (ALT), albumin, glucose, creatinine, uric acid, cholesterol, TG, γ-GT, alkaline phosphatase, total bilirubin, D-Bil, BUN, TP, GLO, HBsAg and Anti-HCV.
* Normal hematology results (within normal range or considered not clinically significant by the investigator) including: hemoglobin, hematocrit, WBC count with differential, RBC count and platelet count.
* Normal urinalysis results (within normal range or considered not clinically significant by the investigator) including: glucose, protein, RBC, WBC, epith, casts and bacteria.
* Female subject who is using adequate contraception since last menstruation and no plan for conception during the study
* Female subject who is non-lactating
* Female subject who has negative pregnancy test (urine) within 14 days prior to the study
* Informed consent form signed

Exclusion Criteria:

* A recent history of drug or alcohol abuse
* Medical history of allergic asthma or sensitivity to analogous product
* A clinically significant illness within the past 4 weeks.
* Evidence of any clinical significant renal, cardiovascular, hepatic, hematopoetic, neurological, pulmonary or gastrointestinal pathology within the past 4 weeks.
* Ongoing peptic ulcer and constipation.
* Planed vaccination during the time course of the study.
* Participation of any clinical investigation during the last 60 days.
* Regular use of any medication during the last 4 weeks.
* Single use of any medication during the last one week.
* Blood donation of more than 500 mL within the past 12 weeks.
* Individuals are judged by the investigators or co-investigator to be undesirable as subjects.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Choo-Aun Neoh, Principal Investigator — PingTung Christian Hospital
Locations (1):
- PingTung Christian Hospital, Pingtung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Hsiao G, Shen MY, Lin KH, Lan MH, Wu LY, Chou DS, Lin CH, Su CH, Sheu JR. Antioxidative and hepatoprotective effects of Antrodia camphorata extract. J Agric Food Chem. 2003 May 21;51(11):3302-8. doi: 10.1021/jf021159t. PMID 12744658

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-one (31) healthy adult subjects enrolled the study. The study period was a continuous 90-day. Each subject received GD Antrodia Camphorata (as three 500 mg capsules) at 7:30 and 19:30 for continuous 90- day.
Pre-assignment Details: One participant didn't continue on the trial by his own will.
Period: Overall Study
Arm/Group | GD Antrodia Camphorata
Started | 31
Completed | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Laboratory measurements, including serum glutamic oxaloacetate transaminase (SGOT), serum glutamic pyruvate transaminase (SGPT), albumin, glucose, creatinine, uric acid, cholesterol, Triglycerides (TG), r-glutamyl transpeptidase(r-GT), alkaline phosphatase, total bilirubin, Direct- bilirubin (D-Bil), BUN, Total protein (TP), Globulin (GLO).
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 20
Region of Enrollment [Number; unit: participants]
  Taiwan | 31
Serum glutamic oxaloacetic transaminase SGOT (AST) [Mean (Standard Deviation); unit: U/L] — Blood was sampled from an antecubital vein of the forearm for the laboratory measurement at 07:30 in the morning. Qualified medical personnel will attend the whole study. No smoking, alcohol and caffeine consumption will be permitted for at least 48 hours before and during the study.
  U/L | 16.74 (3.95)
Serum glutamic pyruvate transaminase, SGPT (ALT) [Mean (Standard Deviation); unit: U/L] — Subjects would fast for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  U/L | 17.32 (9.03)
Triglycerides (TG) [Mean (Standard Deviation); unit: mg/dL] — Subjects would fast for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 in the morning. Qualified medical personnel will attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  mg/dL | 75.19 (35.16)
Total protein [Mean (Standard Deviation); unit: g/dL] — The total protein test measures the total amount of two classes of proteins in the blood, albumin and globulin. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 am. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  g/dL | 6.88 (0.32)
Uric acid [Mean (Standard Deviation); unit: mg/dL] — Subjects would fast for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 in the morning.
  mg/dL | 5.79 (1.13)
Albumin [Mean (Standard Deviation); unit: g/dL] — Subjects would fast for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 in the morning. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  g/dL | 4.47 (0.16)
Alkaline phosphatase [Mean (Standard Deviation); unit: U/L] — Subjects would fast for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 in the morning. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  U/L | 52.06 (13.18)
Direct bilirubin [Mean (Standard Deviation); unit: mg/dL] — Bilirubin is brownish yellow substance found in bile. It's produced when the liver breaks down old red blood cells. Bilirubin circulates in the bloodstream in two forms: indirect and direct bilirubin. Direct bilirubin is made by the liver from indirect form. This test can be used to check the liver function. Subjects would fast for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement.
  mg/dL | 0.16 (0.06)
Total bilirubin [Mean (Standard Deviation); unit: mg/dL] — Total bilirubin is referred to the sum of direct bilirubin and indirect bilirubin. Direct bilirubin is water- soluble form, made by the liver. Indirect bilirubin is not soluble in water due to the intramolecular hydrogen bond. Indirect bilirubin circulates in plasma. Total bilirubin test can be used to check liver function and haemolytic disease. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 in the morning. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  mg/dL | 0.80 (0.28)
BUN [Mean (Standard Deviation); unit: mg/dL] — Subjects fasted for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 am. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  mg/dL | 10.70 (2.53)
Cholesterol [Mean (Standard Deviation); unit: mg/dL] — Subjects fasted for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 in the morning. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  mg/dL | 169.10 (27.05)
Creatinine [Mean (Standard Deviation); unit: mg/dL] — Subjects fasted for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 am. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  mg/dL | 0.78 (0.15)
Globulin [Mean (Standard Deviation); unit: g/dL] — Globulin proteins include enzymes, antibodies and more than 500 other proteins. Subjects fasted for 8 hours prior to study product administration at 7:30 am in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement at 7:30 in the morning. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  g/dL | 2.41 (0.32)
r-glutamyl transpeptidase (r-GT) [Mean (Standard Deviation); unit: U/L] — Subjects would fast for 8 hours prior to study product administration at 7:30 in the morning. Blood would be sampled from an antecubital vein of the forearm for the laboratory measurement. Qualified medical personnel would attend the whole study. No smoking, alcohol and caffeine consumption would be permitted for at least 48 hours before and during the study.
  U/L | 14.90 (6.85)

OUTCOME MEASURES:

1. Primary Outcome: Serum Glutamic Oxaloacetic Transaminase (AST/SGOT)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
U/L | 21.48 (6.43)

2. Primary Outcome: Serum Glutamic Pyruvate Transaminase (ALT/SGPT)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
U/L | 21.94 (10.10)

3. Primary Outcome: Triglycerides (TG)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 56.39 (23.17)

4. Primary Outcome: Total Protein
Description: The total protein test measures the total amount of two classes of proteins in the blood, albumin and globulin.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
g/dL | 7.25 (0.34)

5. Primary Outcome: Uric Acid
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 5.47 (1.25)

6. Primary Outcome: Albumin
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
g/dL | 4.74 (0.20)

7. Primary Outcome: Alkaline Phosphatase
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
U/L | 55.81 (14.33)

8. Primary Outcome: Direct Bilirubin
Description: Direct bilirubin is referred to as conjugated bilirubin, which is water-soluble. It's taken up by the liver cells and conjugated to form the water-soluble bilirubin diglucuronide. It's used to diagnose and/or monitor liver diseases, such as cirrhosis, hepatitis or gallstones. If direct bilirubin is elevated more than unconjugated bilirubin, there's typically a problem associated with decreased elimination of bilirubin by the liver cells.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 0.10 (0.07)

9. Primary Outcome: Total Bilirubin
Description: Bilirubin is released into the blood when red blood cells break down. The liver uses bilirubin to make bile. Normally there is only a small amount of bilirubin in the blood. High levels may be caused by liver or blood problems.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 0.73 (0.32)

10. Primary Outcome: BUN
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 9.32 (2.49)

11. Primary Outcome: Cholesterol
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 173.13 (28.09)

12. Primary Outcome: Creatinine
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 0.84 (0.16)

13. Primary Outcome: Globulin
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
g/dL | 2.51 (0.29)

14. Primary Outcome: Glucose
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
mg/dL | 80.13 (6.13)

15. Primary Outcome: R-glutamyl Transpeptidase (r-GT)
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | GD Antrodia Camphorata
Number analyzed (Participants) | 31
U/L | 17.42 (7.76)

ADVERSE EVENTS:
Arm/Group | GD Antrodia Camphorata
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No